CLINICAL TRIAL: NCT03471832
Title: Clinical Evaluation of CooperVision MyDay Lenses
Brief Title: Clinical Evaluation of Stenfilcon A Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JP-MKTG-201709_02
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This will be a non-dispensing, randomized, contralateral study comparing a test lens against the appropriate control lens.
Who Masked: Participant
Masking Description: Each subject will be masked as to which lens is worn on each eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- stenfilcon A lens (Experimental): MyDay contact lens
  Interventions: Device: stenfilcon A lens
- narafilcon A lens (Active Comparator): 1-Day Acuvue TruEye
  Interventions: Device: narafilcon A lens

INTERVENTIONS:
Device: stenfilcon A lens — contact lens
  Other Names: MyDay, test
  Arms: stenfilcon A lens
Device: narafilcon A lens — contact lens
  Other Names: 1-day Acuvue TruEye, control
  Arms: narafilcon A lens

SUMMARY:
This study is to evaluate the fitting performance of stenfilcon A contact lens (test) compared to narafilcon A contact lens (control).

DETAILED DESCRIPTION:
This study is to evaluate the fitting performance of stenfilcon A contact lens (test) compared to narafilcon A contact lens (control) over 3 hour of wear time in a Japanese population.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is Japanese
* Has had a self-reported oculo-visual examination in the last two years.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the informed consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
* Currently wears soft contact lenses.
* Has clear corneas and no active ocular disease.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kodama, MD, PhD, Principal Investigator — Kodama Eye Clinic
Locations (4):
- Japan (4):
  - Shioya Eye Clinic, Fukushima, Fukushima
  - Kodama Eye Clinic, Terada, Kyoto
  - Itoi Eye Clinic, Shibuya City, Tokyo
  - Ueda Eye Clinic, Shimonoseki, Yamaguchi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Stenfilcon A Lens: Subjects were randomized to wear stenfilcon A lens and narafilcon A lens in this contralateral, non-dispensing study.
  stenfilcon A lens: contact lens
- Narafilcon A Lens: Subjects were randomized to wear narafilcon A lens and stenfilcon A lens in this contralateral, non-dispensing study.
  narafilcon A lens: contact lens
Period: Overall Study
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Started | 40; 40 Eyes | 40; 40 Eyes
Completed | 40; 40 Eyes | 40; 40 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 40

OUTCOME MEASURES:

1. Primary Outcome: Lens Movement
Description: Movement of lens after blink: (Categories = Tight, Slightly tight, Optimum, Slightly loose, Loose)
Time Frame: 5 minutes
Measure: Number; unit: Number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
Number of eyes
  Tight | 0 | 0
  Slightly tight | 0 | 3
  Optimum | 30 | 30
  Slightly Loose | 10 | 7
  Loose | 0 | 0

2. Primary Outcome: Lens Movement
Description: Movement of lens after blink: (Categories = Tight, Slightly tight, Optimum, Slightly loose, Loose)
Time Frame: 3hrs
Measure: Number; unit: Number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
Number of eyes
  Tight | 0 | 0
  Slightly tight | 5 | 11
  Optimum | 32 | 26
  Slightly Loose | 3 | 3
  Loose | 0 | 0

3. Primary Outcome: Horizontal Lens Centration
Description: Centration of lens horizontally: (Grades = Temporal, Slightly temporal, Centered, Slightly Nasal, Nasal)
Time Frame: 5 minutes
Measure: Number; unit: Number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
Number of eyes
  Temporal | 0 | 0
  Slightly temporal | 4 | 8
  Center | 36 | 32
  Slightly nasal | 0 | 0
  Nasal | 0 | 0

4. Primary Outcome: Horizontal Lens Centration
Description: Centration of lens horizontally: (Grades = Temporal, Slightly temporal, Centered, Slightly Nasal, Nasal)
Time Frame: 3hrs
Measure: Number; unit: number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
number of eyes
  Temporal | 0 | 0
  Slightly temporal | 1 | 8
  Center | 39 | 32
  Slightly nasal | 0 | 0
  Nasal | 0 | 0

5. Primary Outcome: Vertical Lens Centration
Description: Centration of lens horizontally: (Grades = Superior, Slightly superior, Center, Slightly inferior, Inferior)
Time Frame: 5 minutes
Measure: Number; unit: Number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
Number of eyes
  Superior | 0 | 0
  Slightly superior | 3 | 10
  Center | 35 | 27
  Slightly inferior | 2 | 3
  Inferior | 0 | 0

6. Primary Outcome: Vertical Lens Centration
Description: Centration of lens horizontally: (Grades = Superior, Slightly superior, Centered, Slightly inferior, Inferior)
Time Frame: 3hrs
Measure: Number; unit: Count of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
Count of eyes
  Superior | 0 | 0
  Slightly superior | 1 | 6
  Center | 39 | 28
  Slightly inferior | 0 | 6
  Inferior | 0 | 0

7. Primary Outcome: Corneal Coverage
Description: Does lens cover the cornea: (Yes, No)
Time Frame: 5 minutes
Measure: Number; unit: number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
number of eyes
  Yes | 40 | 40
  No | 0 | 0

8. Primary Outcome: Corneal Coverage
Description: Does lens cover the cornea: (Yes, No)
Time Frame: 3hrs
Measure: Number; unit: number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
number of eyes
  Yes | 40 | 40
  No | 0 | 0

9. Primary Outcome: Lens Lag
Description: Movement after looking right and left: (Grades = Move along with cornea, slight delay, delay)
Time Frame: 5 minutes
Measure: Number; unit: number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
number of eyes
  Move along with cornea | 35 | 34
  Slightly Delay | 3 | 5
  Delay | 2 | 1

10. Primary Outcome: Lens Lag
Description: Movement after looking right and left: (Grades = Move along with cornea, slight delay, delay)
Time Frame: 3hrs
Measure: Number; unit: number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
number of eyes
  Move along with cornea | 39 | 36
  Slightly Delay | 1 | 4
  Delay | 0 | 0

11. Primary Outcome: Overall Fitting Performance
Description: Lens fit performance: (Grades: Optimum, Good, Acceptable, Unacceptable)
Time Frame: 5 minutes
Measure: Number; unit: number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
number of eyes
  Optimum | 30 | 25
  Good | 8 | 11
  Acceptable | 2 | 4
  Unacceptable | 0 | 0

12. Primary Outcome: Overall Fitting Performance
Description: Lens fit performance: (Grades: Optimum, Good, Acceptable, Unacceptable)
Time Frame: 3hrs
Measure: Number; unit: number of eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
number of eyes
  Optimum | 32 | 22
  Good | 6 | 14
  Acceptable | 2 | 4
  Unacceptable | 0 | 0

13. Primary Outcome: Investigator Fit Preference
Description: Lens fit preference: (Grades: Prefer stenfilcon A strongly, Prefer stenfilcon A slightly, Either, Prefer narafilcon A slightly, Prefer narafilcon A strongly)
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study - Investigator Fitting Preference: Subjects were randomized to wear stenfilcon A lens and narafilcon A lens in this contralateral, non-dispensing study.
  stenfilcon A lens: contact lens narafilcon A lens: contact lens
Arm/Group | Overall Study - Investigator Fitting Preference
Number analyzed (Participants) | 40
Participants
  Prefer stenfilcon A strongly | 5
  Prefer stenfilcon A slightly | 6
  Either | 24
  Prefer narafilcon A slightly | 4
  Prefer narafilcon A strongly | 1

14. Primary Outcome: Investigator Fit Preference
Description: as for outcome 13
Time Frame: 3hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study - Investigator Fitting Preference
Number analyzed (Participants) | 40
Participants
  Prefer stenfilcon A strongly | 5
  Prefer stenfilcon A slightly | 12
  Either | 17
  Prefer narafilcon A slightly | 6
  Prefer narafilcon A strongly | 0

15. Secondary Outcome: Comfort
Description: Subjective comfort: (on a scale of 0-10, 0 (Uncomfortable) - 10 (Comfortable))
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 8.1 (2.0) | 8.1 (1.9)

16. Secondary Outcome: Comfort
Description: Subjective comfort: (on a scale of 0-10, 0 (Uncomfortable) - 10 (Comfortable))
Time Frame: 5 Minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 8.2 (2.2) | 8.2 (1.9)

17. Secondary Outcome: Comfort
Description: Subjective comfort: (on a scale of 0-10, 0 (Uncomfortable) - 10 (Comfortable))
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 8.2 (2.3) | 8.4 (2.2)

18. Secondary Outcome: Dryness
Description: Subjective dryness: (on a scale of 0-10, 0 (Dry) - 10 (Not dry))
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 9.3 (1.2) | 8.1 (1.9)

19. Secondary Outcome: Dryness
Description: Subjective dryness: (on a scale of 0-10, 0 (Dry) - 10 (Not dry))
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 9.1 (1.5) | 8.2 (1.9)

20. Secondary Outcome: Dryness
Description: Subjective dryness: (on a scale of 0-10, 0 (Dry) - 10 (Not dry))
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 8.5 (1.9) | 8.4 (2.2)

21. Secondary Outcome: Stinging/Burning
Description: Subjective stinging/burning sensation: (on a scale of 0-10, 0 (Cannot wear) - 10 (No Stinging/Burning))
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 9.5 (1.2) | 8.8 (2.3)

22. Secondary Outcome: Stinging/Burning
Description: Subjective stinging/burning sensation: (on a scale of 0-10, 0 (Cannot wear) - 10 (No Stinging/Burning))
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 9.8 (0.7) | 9.0 (1.8)

23. Secondary Outcome: Stinging/Burning
Description: Subjective stinging/burning sensation: (on a scale of 0-10, 0 (Cannot wear) - 10 (No Stinging/Burning))
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 9.6 (1.0) | 9.6 (0.9)

24. Secondary Outcome: Edge/Lens Awareness
Description: Subjective edge/lens awareness: (on a scale of 0-10, 0 (Cannot wear) - 10 (No edge awareness))
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 9.0 (2.0) | 9.4 (1.6)

25. Secondary Outcome: Edge/Lens Awareness
Description: Subjective edge/lens awareness: (on a scale of 0-10, 0 (Cannot wear) - 10 (No edge awareness))
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 8.9 (1.9) | 9.1 (1.6)

26. Secondary Outcome: Edge/Lens Awareness
Description: Subjective edge/lens awareness: (on a scale of 0-10, 0 (Cannot wear) - 10 (No edge awareness))
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
Number analyzed (Participants) | 40 | 40
Number analyzed (Eyes) | 40 | 40
units on a scale | 8.7 (2.4) | 9.2 (1.8)

27. Secondary Outcome: Subjective Lens Preference
Description: Lens preference (stenfilcon A, Either, Neither, narafilcon A)
Time Frame: Baseline
Population: One subject data was excluded as the subjective lens preference was answered only after 3 hours of lens wear.
Measure: Count of Participants; unit: Participants
Groups:
- Lens Preference - After Insertion: Subjects were randomized to wear stenfilcon A lens and narafilcon A lens in this contralateral, non-dispensing study.
  stenfilcon A lens: contact lens
Arm/Group | Lens Preference - After Insertion
Number analyzed (Participants) | 39
Participants
  Prefer stenfilcon A | 14
  Either | 13
  Neither | 1
  Prefer narafilcon A | 11

28. Secondary Outcome: Subjective Lens Preference
Description: Lens preference (stenfilcon A, Either, Neither, narafilcon A)
Time Frame: 5 minutes
Population: One subject data was excluded as the subjective lens preference was answered only after 3 hours of lens wear.
Measure: Count of Participants; unit: Participants
Arm/Group | Lens Preference - After Insertion
Number analyzed (Participants) | 39
Participants
  Prefer stenfilcon A | 13
  Either | 14
  Neither | 2
  Prefer narafilcon A | 10

29. Secondary Outcome: Subjective Lens Preference
Description: Lens preference (stenfilcon A, Either, Neither, narafilcon A)
Time Frame: 3 hours
Population: One subject data was excluded as the subjective lens preference was answered only after 3 hours of lens wear.
Measure: Count of Participants; unit: Participants
Arm/Group | Lens Preference - After Insertion
Number analyzed (Participants) | 39
Participants
  Prefer stenfilcon A | 12
  Either | 18
  Neither | 1
  Prefer narafilcon A | 9

ADVERSE EVENTS:
Time Frame: From insertion over three hours of lens wear
Arm/Group | Stenfilcon A Lens | Narafilcon A Lens
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT03471832/Prot_SAP_000.pdf